CLINICAL TRIAL: NCT05108181
Title: Influence of Muscle Typology and Training Frequency on Chronic Strength Training Adaptations
Brief Title: Muscle Typology and Strength Training Adaptations
Acronym: MT-ST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BC-10253
Record Dates: First submitted 2021-10-12; First posted 2021-11-04 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Muscle Fiber Type; Exercise; Training Frequency
Keywords: Strength training; Muscle typology
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All participants will receive the same training intervention but the subjects are divided into two groups based on an inherent physiological characteristic: the muscle typology. A slow typology group (people with a lot of slow muscle fibers) and a fast typology group (people with a lot of fast muscle fibers). Each participant will train their legs and arms unilateral and one arm and one leg will train two times per week, while the other arm and leg will train three times per week for 9 weeks. The assignment of the limbs to the 3x/week condition and the 2x/week condition is randomized. The training outcomes of the two groups will be compared as well as the within subject differences between training two times per week or training 3 times per week.
Who Masked: Participant
Masking Description: The participants don't know their muscle typology during the study. All participants do the same training intervention, no drugs are taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow muscle typology group (Active Comparator): The participants receive the same exercise training intervention, but they are divided in two groups: a slow typology group and a fast typology group based on their inherent physiological characteristics: their muscle fiber type.
  Interventions: Other: Muscle typology + exercise training; Other: Muscle typology + training frequency
- Fast muscle typology group (Active Comparator): The participants receive the same exercise training intervention, but they are divided in two groups: a slow typology group and a fast typology group based on their inherent physiological characteristics: their muscle fiber type.
  Interventions: Other: Muscle typology + exercise training; Other: Muscle typology + training frequency

INTERVENTIONS:
Other: Muscle typology + exercise training — Exercise training: Participants perform 9 weeks of strength training at 60% of their 1RM.
Other: Muscle typology + training frequency — Training frequency: leg A and arm A of the participants train 3 times per week, leg B and arm B train 2 times per week.

SUMMARY:
The overall aim of this project is to investigate if the responsiveness to chronic resistance training is dependent on the muscle typology. In a second aim we will investigate the most optimal training frequency for slow-twitchers and fast-twitchers. For the latter we hypothesize that slow-twitchers might cope better with higher frequencies and higher volumes compared to fast-twitchers.

Male and female adult participants (18-45y) will be recruited. The subjects' muscle typology will be non-invasively estimated in the leg muscles by measurement of muscle carnosine using H-MRS. In total 21 subjects (11 slow and 10 fast subjects) will participate. Subjects will be assigned to a whole-body resistance training exercise protocol of 9 weeks in wich arm A and leg A will train 3 times per week and arm B and leg B will train 2 times per week. Before and following the training period, subjects will be subjected to different measurements (fitness level, muscle volume, strength tests, blood sampling, muscle biopsies).

ELIGIBILITY:
Inclusion Criteria:

* Fast or slow muscle typology
* 18 - 45 years old
* no strength training experience

Exclusion Criteria:

* Vegan/vegeterian diet
* Supplement intake
* chronic diseases
* Hypertension,
* Smoking
* Medication use
* Coagulation disorder, infectious diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline muscle volume at 9 weeks | Pre and post the 9 weeks training period
  Muscle volume of the legs and the upper arms - MRI
Change from baseline dynamic muscle strength at 3 weeks | Pre, mid and post 9 weeks training period
  Upper legs and upper arms - strength training devices
Change from baseline dynamic muscle strength at 6 weeks | Pre, mid and post 9 weeks training period
  Upper legs and upper arms - strength training devices
Change from baseline dynamic muscle strength at 9 weeks | Pre, mid and post 9 weeks training period
  Upper legs and upper arms - strength training devices
Change from baseline isometric muscle strength at 9 weeks | Pre and post 9 weeks training period
  Upper legs and upper arms - Biodex
Change in muscle fiber type specific hypertrophy at 9 weeks | Pre and post 9 weeks training period
  Legs - Biopsy (vastus lateralis)

SECONDARY OUTCOMES:
Change of baseline antropometry at 9 weeks | Pre and post 9 weeks training period
  Height, weight, skinfolds
Change of baseline skeletal muscle protein content at 9 weeks | Pre and post 9 weeks training period
  Histochemistry and protein content of markers of relevance for skeletal muscle function
Change of baseline histochemistry at 9 weeks | Pre and post 9 weeks training period
  Histochemistry of markers of relevance for skeletal muscle function
Change from basline fatigue feeling over 9 weeks training period | Assessed every training during the 9 weeks training period
  Number of repetitions during every training, questionnaire (VAS-scale) before every training, RPE after every training
Change from baseline fasting insulin, glucose, cholesterol and triglycerides at 9 weeks | Pre and post 9 weeks training period
  Fasted blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Wim Derave, Principal Investigator — University Ghent
Locations (1):
- Department of Movement and Sports Sciences, Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No